CLINICAL TRIAL: NCT03874143
Title: Clinical Evaluation of the Use of an mHealth Intervention on Quality of Care Provided by Community Health Workers in Southwest Niger
Brief Title: Clinical Evaluation of the Use of an mHealth Intervention on Quality of Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Vision Canada (Other)
Collaborators: World Health Organization (Other); Ministry of Public Health Niger (Unknown); Toronto Metropolitan University (Other); Global Affairs Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 001
Record Dates: First submitted 2019-02-26; First posted 2019-03-14 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Malaria; Diarrhea; Acute Respiratory Infection
MeSH Terms: conditions — Malaria; Diarrhea | interventions — Quality of Health Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RCom equipped with a smartphone (Experimental)
  Interventions: Other: mHealth Intervention for Quality of Care
- RCom with paper-based system (No Intervention)

INTERVENTIONS:
Other: mHealth Intervention for Quality of Care — Does use of a specially equipped smartphone make a difference in the diagnosis and treatment by RCom of malaria, pneumonia and diarrhea in children aged 2 to 59 months
  Arms: RCom equipped with a smartphone

SUMMARY:
Under the World Health Organization's (WHO) integrated community case management (iCCM) Rapid Access Expansion Program (RAcE), World Vision Niger and Canada supported the Niger Ministry of Public Health to implement iCCM in four health districts in Niger in 2013. Community health workers (CHWs), known as Relais Communautaire (RCom), were deployed in their communities to diagnose and treat children under five years of age presenting with diarrhea, malaria and pneumonia and refer children with severe illness to the higher-level facilities. Two of the districts piloted RCom using smartphones equipped with an application to support quality case management and provide good timely clinical data. A two-arm cluster randomized trial assessed the impact of use of the mHealth application mainly on quality of care (QoC), but also on motivation, retention and supervision

ELIGIBILITY:
Inclusion Criteria:

* children presenting symptoms of illness

Exclusion Criteria:

-

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 520 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Quality of Care (QoC) provided by RCom | 30 weeks
  The maximum QoC score was 31 points; the score was weighted with two-thirds of the score allocated to screening questions and correct identification of the danger signs and signs/symptoms of serious conditions A perfect score was achieved when RComs asked all 10 health screening questions and correctly classified 4 major danger signs and 6 serious symptoms, made appropriate referral, and provided advice to caregivers.